CLINICAL TRIAL: NCT04808726
Title: Effect of Breastfeeding Training on Breastfeeding Success Using The Teach Back Method: Randomized Controlled Study
Brief Title: Breastfeeding Success Using The Teach Back Method
Acronym: BSUTTBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Arzu KUL UÇTU, Ph.D.Assistant Professor, Bozok University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BozokU
Record Dates: First submitted 2019-08-05; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Teach-Back Communication; Breastfeeding
Keywords: breastfeeding; midwife; teach-back; Self-Efficacy; Breastfeeding Support
MeSH Terms: conditions — Teach-Back Communication; Breast Feeding

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental research design
Masking Description: The randomization process was created by a neutral researcher who was not involved in the study. The women were not informed about the groups they were in. Single blind was provided in the study by knowing which group they would be in by the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control Group (Other): standard breastfeeding education and counseling service to another group
  Interventions: Behavioral: Teach Back Method

INTERVENTIONS:
Behavioral: Teach Back Method — Effect of Breastfeeding Training on Breastfeeding Success Using The Teach Back Method: Randomized Controlled Study
  Other Names: Breastfeeding Support

SUMMARY:
Objective: The aim of this study was to evaluate the effect of breastfeeding education on breastfeeding success by using the method described in the information. In addition, it is aimed that the teach-back method will be gained to our national literature and be a guide to the health professionals in their applications in our country.

Materials and Methods: The study was conducted with randomized controlled experimental research design. The study was conducted between 15 January and 15 December 2018 in Yozgat City Hospital and Family Health Centers where women are affiliated. The study was performed with 80 primiparous women as intervention (n: 40) and control (n: 40) groups. The teach-back method is applied to the intervention group and standard education method is applied to the control group to give breastfeeding education. In the study, data collection tools, introductory information collection form, LATCH Breastfeeding Diagnostic and Evaluation Scale, Breastfeeding Self-Efficacy Short Form Scale were used. The data were collected between the first 24 hours, 2nd and 5th days postpartum, on the 13th and 15th days and the 30th and 40th days. Independent t-test, multivariate and one-way analysis of variance, Bonferroni-matched paired t-test were used to evaluate the data.

.

DETAILED DESCRIPTION:
It is important to plan and implement initiatives to increase breast milk intake with numerous benefits in terms of mother and baby health. It is stated that these interventions initiate breastfeeding in the early period and increase the rates of breastfeeding. It is stated that breastfeeding success and duration are influenced by many factors such as health status of the baby, mother's demographic characteristics, psychological factors, social support and professional support. It is emphasized that breastfeeding self-efficacy is the most important factor in breastfeeding to maintain healthy and sufficient time. Breastfeeding self-efficacy refers to the full effort of the mother in order to breastfeed her baby, whether she is emotionally ready to breastfeed, and her thoughts on breastfeeding. Demonstrates the ability of the mother to cope with the difficulties she will face in the breastfeeding process.

Determining the factors affecting the continuation of breastfeeding from the prenatal period, breastfeeding support and training against possible risks increase breastfeeding performance. The global vurgulan Baby Friendly Hospital ır application and the Barcelona Declaration of 2001 emphasize that every woman should be encouraged to be informed about breastfeeding and to encourage breastfeeding. Within the framework of these internationally accepted contracts, different educational practices have been introduced to start and sustain breastfeeding.

Breastfeeding trainings can be given by all health personnel such as midwives, nurses, physicians or dieticians. In addition to this, breast-feeding training is offered to individuals who serve voluntarily. Trainings can be carried out individually or in support groups. The planning, implementation and follow-up of breastfeeding education should be carried out periodically. Within the framework of the training programs to be implemented, it is emphasized that mothers should take more role in their health audits in order to maintain breastfeeding self-efficacy and to maintain well-being. The development of breastfeeding self-efficacy is influenced by many variables. However, it is stated that the mother will increase her self-care skills and increase her proportionality with the encouragement of her baby to be breastfed. In order to improve the self-care of the postpartum mother and to increase her participation in health, various theory and approach models are used. Among these, Dorote Orem's Self-Care Theory, Health Belief Model, and Teach-Back Method, which is recently described as a communication technique, are frequently recommended.

Using Teach-Back method, health personnel service management and service service guiding design in the framework of the framework, to use the time effectively, to provide a more professional way to provide service delivery. Health institutions are expected to reduce health care costs by reducing returns. The unconditional fact that individuals are given al understood liği means that they are learned with their own sentences and the use of the subject in this regard expects to reduce the complications and take the level of experience and experience when the investigators can go to breastfeeding after the birth of one of our members. Also the use of usulem; It will be possible to supervise the understanding of the transferred information in a systematic, space for the education and services that will be given at the end of birth. Health literacy and health-related quality of life in this method of learning.

Purpose of the research The aim of this study is to evaluate the effect of breastfeeding education on breastfeeding success. In addition, the method of telling the learned method is aimed to be recognized in our country and to guide health professionals in health services.

Research Hypotheses H0: Using the Teach-Back method, breastfeeding education has no effect on breastfeeding success.

H1: The teaching of breastfeeding by using the Teach-Back method has an effect on the success of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Know reading
* Primiparity
* Term and healthy birth
* Having a healthy newborn
* Vaginal delivery

Exclusion Criteria:

* Not knowing Turkish
* Multiparousness
* Early childbirth
* The health status of the newborn is not good
* Caesarean delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-03-24 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
LATCH Breastfeeding Diagnosis and Evaluation Scale | 2 months
  LATCH Breastfeeding Diagnosis and Evaluation Scale provides a systematic and comprehensive method for obtaining information on themother's breastfeeding capabilities. The system assigns anumerical score of 0, 1 or 2 to ﬁve major elements of breast-feeding. The letters of the acronym LATCH denote the areasof the charting system, as follows: (L) for how well the babyattaches to the breast, (A) for the number of swallows, (T) forthe nipple type, (C) for the maternal comfort grade and (H)for the amount of assistance that the mother requires whenholding her baby to her breast. The total score obtained fromthe evaluation of breastfeeding is 10; a total score that isbelow 10 indicates that the mother requires support
Postpartum Breastfeeding Self-Efficacy Scale Short Form | 2 months
  Postpartum Breastfeeding Self-Efficacy Scale Short Form has14 items. The 14 items in the BSES-SFcontain statements about coping with and managing breast-feeding as well as feelings about breastfeeding skills. Thetotal scores to be obtained from the BSES-SF range from 14-70; a higher average score denotes a higher level of breast-feeding self-efﬁcacy
Personal information form | 2 months
  socio-demographic and personal characteristics questions related to birth, postpartum period and breastfeeding

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat City Hospital, Yozgat, City Center, Turkey (Türkiye)

REFERENCES:
- [Derived] Kul Uctu A, Ozerdogan N. Effect of teach-back method on breastfeeding success: A single blind randomized controlled study. Health Care Women Int. 2023 Mar;44(3):314-327. doi: 10.1080/07399332.2021.2021915. Epub 2022 Feb 17. PMID 35175908

DOCUMENTS (3):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04808726/Prot_SAP_ICF_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04808726/SAP_001.pdf
  • Informed Consent Form: Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04808726/ICF_002.pdf